CLINICAL TRIAL: NCT03309150
Title: A Rollover Study to Provide Continued Treatment With M6620
Brief Title: ATRi Transition Rollover Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS201923-0007; 2017-002354-37 (EudraCT Number)
Record Dates: First submitted 2017-10-10; First posted 2017-10-13 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-10

CONDITIONS: Advanced Stage Solid Tumors
Keywords: Ataxia telangiectasia mutated and Rad3-related protein inhibitor (ATRi); M6620; Solid tumors
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies | interventions — berzosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Part A1: Berzosertib (Experimental)
  Interventions: Drug: Berzosertib

INTERVENTIONS:
Drug: Berzosertib — Participants received intravenous infusion of Berzosertib at a dose of 126 milligrams (mg) on Days 1, 8 and 15 until disease progression or unacceptable toxicity occurred.
  Other Names: M6620

SUMMARY:
The main purpose of the study was to monitor the safety of participant receiving long-term treatment of Berzosertib as monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants ongoing treatment in Vertex study VX13-970-002.
* Participant must be able to understand and provide written informed consent.
* Participant must be willing and able to comply with the scheduled visits, treatment plan, lifestyle, laboratory tests, contraceptive guidelines, and other study procedures.

Exclusion Criteria:

* Participants experiencing disease progression or unacceptable toxicity at the time of transition into the this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, United Kingdom

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201923-0007
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant from Part A1 of Study VX13-970-002 (parent study) was transferred to this study to continue receiving berzosertib.
Groups:
- Part A1: Berzosertib: Participants received intravenous infusion of Berzosertib at a dose of 126 milligrams (mg) on Days 1, 8 and 15 until disease progression or unacceptable toxicity occurred.
Period: Overall Study
Arm/Group | Part A1: Berzosertib
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Part A1: Berzosertib
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Race-White | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Treatment Related AEs
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, regardless of causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Treatment-related AEs: reasonably related to the study intervention.
Time Frame: Up to 6 years
Population: Safety analysis set (SAF) included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Berzosertib: Participants received intravenous infusion of Berzosertib at a dose of 126 milligrams (mg) on Days 1, 8 and 15 until disease progression or unacceptable toxicity occurred.
Arm/Group | Part 1: Berzosertib
Number analyzed (Participants) | 1
Participants
  AEs | 1
  Treatment related AEs | 0

ADVERSE EVENTS:
Time Frame: Up to 6 years
Arm/Group | Part A1: Berzosertib
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A1: Berzosertib (N=1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (3)
Oral candidiasis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT03309150/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/50/NCT03309150/SAP_001.pdf